CLINICAL TRIAL: NCT06771544
Title: Metronomic Cyclophosphamide With Pembrolizumab in Checkpoint Inhibitor Refractory Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Warren Chow, HS Clinical Professor and Associate Director for Clinical Science, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6168; UCI 22-49 (Other: UCI CFCCC)
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-01

CONDITIONS: Melanoma; Melanoma Stage III; Melanoma (Skin); Melanoma Stage IV
Keywords: Melanoma; Melanoma, Stage III; Skin; Melanoma, Stage IV; Pembrolizumab; Cyclophosphamide
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab + Cyclophosphamide (Experimental): Pembrolizumab 200mg IV every 21 days or 400 mg IV every 42 days Cyclophosphamide 50mg PO daily on days 1-14 every 21 days for melanoma patients
  Interventions: Drug: Pembrolizumab; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Pembrolizumab — Given IV
Drug: Cyclophosphamide — Given PO

SUMMARY:
This is a phase 2, single-arm, open label clinical trial determining efficacy of Cyclophosphamide and Pembrolizumab in subjects with melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of signing informed consent form (ICF)
* Patients must have unresectable Stage III or Stage IV non-ocular melanoma per American Joint Committee on Cancer 8th Edition Staging Criteria not amenable to local therapy
* Participants must have measurable disease by RECIST v1.1 criteria as assessed by investigator/ radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been shown in such lesions.
* Participants must have Eastern Cooperative Group (ECOG) performance status score of 0, 1 or 2 at screening visit.
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver, and renal function
* Hemoglobin ≥9.0 g/dL
* Platelets ≥100/mm3
* ANC ≥1.5/mm3
* Creatinine Clearance ≥ 30mL/min Cockcroft-Gault CrCl, mL/min = (140 - age) × (weight, kg) × (0.85 if female) / (72 × Cr, mg/dL).
* AST and ALT less than 3 times the Upper Limit of Normal or less than 5 times the Upper Limit of normal with liver metastases. T Bilirubin < 3.1 mg/dL.
* Has progressed on a prior PD-1/PD-L1 treatment
* Recovered from toxicities of pembrolizumab to Grade ≤1, excluding endocrine toxicities
* Prior Receipt of PD-1/PD-L1 therapy within 9 weeks prior to the first dose of the investigational therapy.
* Women of childbearing potential must have had a negative pregnancy test performed within 7 days prior to the start of treatment
* Females of childbearing potential and males must be willing and able to use an adequate method of contraception to avoid pregnancy for the duration of the study.
* Male and female participants of childbearing potential who are sexually active with a non-sterilized partner must agree to use highly effective methods of birth control from the trial screening date until 3 months after the final dose of study intervention; cessation of birth control after this point shall be discussed with a responsible physician.
* Pregnant or lactating women are prohibited from enrolling in this study.
* Male participants are not allowed to donate sperm from the time of enrollment until 6 months after administration of study interventions.

Exclusion Criteria:

* Participants with a diagnosis of ocular or metastatic uveal melanoma
* Participants with a history of a malignant disease other than those being treated in this study. The following exceptions are permitted:
* Malignancies that were treated curatively and have not recurred within 2 years. Shorter intervals can be considered after discussion with the Principal Investigator.
* Completely resected basal cell and squamous cell skin cancers.
* Any malignancy considered to be indolent and that has never required therapy, such as chronic lymphocytic leukemia.
* Completely resected carcinoma in situ of any type
* Participants ineligible to be retreated with pembrolizumab due to a treatment-related AE while on a prior anti-PD(L)-1 regimen that led to discontinuation of that prior therapy and would thus prevent retreatment or with an immune-related adverse event (irAE) of grade 3 or greater
* Participants with known untreated or symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis. NOTE: Participants with previously treated brain metastases may participate provided ALL of the following apply:
* Treated CNS lesions are radiographically stable (without evidence of progression for ≥ 28 days prior to the first dose of study intervention) after intervention (eg, surgery and/or radiation).
* Neurologically stable and on stable dose of ≤ 10mg of prednisone equivalent steroids for at least 7 days prior to the first dose of study intervention.
* Any prior investigational or standard cancer therapy, with exception of PD-1/PD-L1 (includes nivolumab + Relatlimab) therapy, chemotherapy or radiation within 6-9 weeks of the first dose of the investigational therapy (see Inclusion Criteria)
* Presence of B-RAF driver mutation without prior receipt of BRAF +/- MEK inhibitors, unless patient declines BRAF +/-MEK inhibition for any reason or is unable to tolerate BRAF and/or MEK inhibitors.
* Participants with a known history of chronic viral infections as indicated below. If patients do not have a known history, testing is not required during the screening period to confirm the patient has an active infection.
* Known HBV infection defined as hepatitis B surface antigen reactive. NOTE: Participants with HBV infection on stable anti-viral therapy for > 4 weeks prior to the planned first study intervention and viral load confirmed as undetectable during Screening may be eligible.
* Known active HCV infection defined as detectable HCV RNA (qualitative) infection. NOTE: History of HCV is not exclusionary if participant has received curative treatment and viral load is confirmed as undetectable during Screening.
* Active HIV infection. Those with HIV infections on combination antiretroviral medications with stable CD4 count >200/microliters as measured within screening time period. If the patient does not have a known history of HIV, then testing is not required during screening to confirm presence or absence of HIV.
* Positive serum pregnancy test
* Participants with out-of-range screening laboratory values as defined below. NOTE: Hematology evaluations must be performed >7 days from any blood transfusion. Or blood product transfusion or from any dose of hematologic growth factor.
* Glomerular filtration rate (calculated using the Chronic Kidney Disease Epidemiology Collaboration formula) < 30 mL/min
* Total bilirubin > 1.5 × ULN; participants with Gilbert's syndrome are excluded if total bilirubin > 3.0 × ULN; or direct bilirubin > 1.5 × ULN
* Albumin < 3.0 g/dL
* Absolute lymphocyte count < 0.5 × 10^9/L
* Participants with a history of allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by RECIST v1.1 | Up to 3 years
  Sum of Complete Response (CR) and Partial Response (PR) by RECIST v 1.1. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1): Complete Response (CR) is defined as the disappearance of all target lesions; Partial Response (PR) is defined as a 30% decrease in the sum of diameters of target lesions. ORR = CR + PR
Number of Patients with Adverse Events | Up to 3 years
  Number of Patients who received at least one dose of Pembrolizumab with Cyclophosphamide with any reported Adverse Events (AEs) using the CTCAE version 5.0 for reporting of nonhematologic AEs and modified criteria for hematologic AEs.
Number of Patients with Immune Related Adverse Events | Up to 3 years
  Number of Patients who received at least one dose of Pembrolizumab with Cyclophosphamide with reported immune related AEs (irAEs) using the CTCAE version 5.0 for reporting of nonhematologic AEs and modified criteria for hematologic AEs.
Number of Patients who Discontinued Treatment Due to Reported Adverse Events | Up to 3 years
  Number of Patients who received at least one dose of Pembrolizumab with Cyclophosphamide requiring discontinuation of therapy due to reported AEs using the CTCAE version 5.0 for reporting of nonhematologic AEs and modified criteria for hematologic AEs..
Comparative Analysis of Immune Cells | Up to 3 years
  Mean, median, percentage and total counts of immune T cell subsets pre-treatment and after 2 three-week cycles of metronomic cyclophosphamide and pembrolizumab.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by iRECIST | Up to 3 years
  Sum of Complete Response (CR) and Partial Response (PR) by Immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST). Per iRECIST: Immune Complete Response (iCR) is defined the complete disappearance of the tumor and non-tumor lesions; Immune Partial Response (iPR) is defined as a 30% tumor load decrease from baseline; Immune Stable Disease (iSD) is defined as when neither iCR nor iPR apply and there is no tumor progression; Unconfirmed Progressive Disease (iUPD) is defined as a 20% or greater increase in tumor burden or an appearance of a new target or non-target lesion; Confirmed Progressive Disease (iCPD) is defined as an increase of 5mm or greater in target tumor burden, or new target lesion, or any increase in non-target disease; Immune Best overall Response (IBOR) is defined as the best timepoint response recorded from the start to the end of the immunotherapy. ORR based on iRECIST refers to the percentage of patients in a clinical trial who experience a measurable
Clinical Benefit Rate | Up to 3 years
  Complete Response, Partial Response, and >6 months of stable disease as evaluated by RECIST v 1.1 and immune RECIST (iRECIST).
  Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1): Complete Response (CR) is defined as the disappearance of all target lesions; Partial Response (PR) is defined as a 30% decrease in the sum of diameters of target lesions. Stable Disease is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study
Overall Survival | Up to 3 years
  Survival rate of subjects who received at least one dose of Pembrolizumab with Cyclophosphamide
Progression Free Survival | Up to 3 years.
  Survival rate of subjects who received at least one dose of Pembrolizumab with Cyclophosphamide without Progression of their disease.
Duration of Response | Up to 3 years
  Duration of Response of subjects who received at least one dose of Pembrolizumab with Cyclophosphamide

OTHER OUTCOMES:
Comparison of Phenotype and T-Cell Function | Up to 3 years
  Compare the Phenotype of and T-cell Function of Paired Biopsies before and after Investigational Treatment
Comparative Quantitative analysis of T-Cell Repertoire | Up to 3 years
  Comparative Quantitative analysis of T-Cell Repertoire in Paired Biopsies before and after Investigational Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Warren Chow, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No